CLINICAL TRIAL: NCT02055482
Title: A Controlled, Parallel Group, Open-label, Multicenter Extension Study to Investigate Efficacy and Safety of Oral BAY85-3934 and Darbepoetin Alfa Comparator in the Long Term Treatment of Anemia in Pre-dialysis Subjects With Chronic Kidney Disease in Europe and Asia Pacific
Brief Title: Long-term Pre-dialysis Extension in Europe and Asia Pacific
Acronym: DIALOGUE 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15653; 2013-001190-24 (EudraCT Number)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Anemia; Renal Insufficiency, Chronic
Keywords: Anemia on CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY85-3934 (Experimental)
  Interventions: Drug: Molidustat (BAY85-3934)
- Darbepoetin (Active Comparator)
  Interventions: Biological: Darbepoetin

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — BAY85-3934 will be titrated at the scheduled dose control visits to maintain the Hb in the target range of 10.0 to 12.0 g/dL. Available doses include 15, 25, 50, 75, 100, and 150 mg/day OD. Treatment will be for minimum of 6 months to up to a maximum of 36 months.
  Arms: BAY85-3934
Biological: Darbepoetin — Darbepoetin will be administered according to the local label and titrated at the scheduled dose by intravenous injection. Treatment will be for a minimum of 6 months to up to a maximum of 36 months.
  Arms: Darbepoetin

SUMMARY:
Anaemia is a condition in which blood has a lower than normal number of red blood cells. It can also occur if red blood cells do not contain enough haemoglobin, an oxygen carrying part of blood. Anaemia is common in patients with chronic kidney disease. Healthy kidneys produce a hormone called erythropoietin, which stimulates the bone marrow to produce the proper number of red blood cells needed to carry oxygen to vital organs. Chronic kidney disease is a general term that means that the kidneys are not functioning to their full potential. The study drug, BAY85-3934, is being evaluated as a drug to increase the body's ability to produce erythropoietin.

The purpose of this extension study is to find out if the study drug, a tablet taken orally, is safe and effective for the treatment of anaemia associated with chronic kidney disease.

The extension study will enroll up to 240 patients at multiple locations in Europe, Asia and Australia. Patients who participated in Studies 15141 or 15261 may be eligible to take part in the extension study. The study consists of the Haemoglobin (Hb) Stabilisation Phase and the Main Phase. The Hb Stabilisation Phase involves up to 10 study visits scheduled over 16 weeks. The Main Phase will last for at least 6 months and up to a maximum of 36 months, with visits every 4 weeks. During these scheduled visits patients will undergo a number of procedures to confirm efficacy and safety of the study drug, including measurement of heart rate and blood pressure, physical examination, Electrocardiogram and blood/urine sample collection for laboratory tests.

The study will be conducted at 5 hospitals in the UK. Bayer HealthCare AG is funding this research. This study will include subjects who either completed the treatment period in their respective Phase 2 parent study (i.e., Study 15141 or Study 15261) or experienced a stopping event in the fixed dose parent study (Study 15141). As Study 15141 is a double-blind study, subjects will be unblinded as per the Study 15141 protocol prior to entry into the extension study.

ELIGIBILITY:
Inclusion Criteria:

* Men who agree to use adequate contraception when sexually active or women without childbearing potential
* Not on dialysis at study entry
* Serum ferritin levels ≥ 100 μg/L and < 1000 μg/L or transferrin saturation ≥ 20%
* Inclusion criteria for inclusion into the Hb Stabilization (HbS) Phase: Requires Hb stabilization (at 10.0 to 12..0g/dL for a minimum of 4 weeks) as follows: Received BAY 85-3934 and reached a stopping event in Study 15141 or received placebo and reached a stopping event in Study 15141 or completed 16 weeks of treatment with BAY 85-3934 in Study 15141or 15261 but had mean Hb during the evaluation period outside the target range of 10.0 to 12.0 g/dL, or Completed 16 weeks of treatment with placebo in Study 15141 and was re-assessed at 4 weeks after end of study as eligible for Study 15653 (this study)
* Inclusion criteria for inclusion into the Main Phase: Mean Hb concentration of 10.0 to 12.0 g/dL who completed 16 weeks of treatment (BAY85-3934 arm) in Study 15141, or completed 16 weeks of treatment (BAY-3934 or darbepoetin arm)in study 15261 without a dose suspension lasting > 6 consecutive weeks, or mean Hb concentration of 10.0 to 12.0g/dL during the HbS phase of Study 15653 for a minimum of 4 weeks after visit 3.

Exclusion Criteria:

* A scheduled kidney transplant or any other organ transplant within the next 6 months (being on a waiting list does not exclude the subject)
* Red blood cell (RBC) containing transfusion within the 8 weeks before baseline
* Phosphodiesterase type 5 (PDE5) inhibitor (e.g., sildenafil, vardenafil, tadalafil) or nitrates
* Sustained, poorly controlled arterial hypertension or hypotension at baseline, defined as blood pressure ≥ 180/110 mmHg or systolic blood pressure < 95 mmHg, respectively
* Severe rhythm or conduction disorders (e.g., heart rate [HR] < 50 or > 110 bpm, atrial flutter, prolonged QT > 500 msec, second or third degree atrioventricular [AV] block), if not reacted with a pace marker)
* New York Heart Association Class III or IV congestive heart failure
* Severe hepatic insufficiency (defined as alanine aminotransferase [ALT], aspartate aminotransferase [AST]>3x the upper limit of normal [ULN], total bilirubin > 2 mg/dL, or Child Pugh B or C) or active hepatitis, in the investigator's opinion
* An ongoing serious adverse event (SAE) from Study 15141 or Study 15261 that is assessed as related to study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory hemoglobin level from baseline | Baseline up to 36 months
Number of participants with serious adverse events (SAEs) and adjucated adverse events as a measure of safety and tolerability | Up to 36 months
Number of participants with liver function-related AEs including abnormal liver function tests and any hospitalization | Up to 36 months

SECONDARY OUTCOMES:
Time within hemoglobin target range (10.0 to 12.0 g/dL) | Up to 36 months
Duration of treatment exposure | Up to 36 months
Number of subjects requiring titration of dose | Up to 36 months
Change of reticulocyte count from baseline of this study | Baseline up to 36 months
Change of red blood cell count from baseline of this study | Baseline up to 36 months
Change of hematocrit from baseline of this study | Baseline up to 36 months
Change of central laboratory hemoglobin level from baseline of this study | Baseline up to 36 months
Responders in Hb levels | Up to 36 months
Number of subjects meeting specific Hb criteria | Baseline up to 36 months
Number of subjects with Hb values >13 g/dL or having excessive Hb increase | Baseline up to 36 months
Number of participants with non-serious adverse events | Up to 36 months
Change in heart rate (HR) | Up to 36 months
Change in blood pressure (BP) | Up to 36 months
Laboratory abnormalities | Up to 36 months

OTHER OUTCOMES:
Change of reticulocyte count from baseline of study 15141 or 15261 | Baseline up to 36 months
Change of red blood cell count from baseline of study 15141 or 15261 | Baseline up to 36 months
Change of hematocrit from baseline of study 15141 or 15261 | Baseline up to 36 months
Change of central laboratory hemoglobin level from baseline of study 15141 or 15261 | Baseline up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (93):
- Australia (3):
  - Gosford, New South Wales
  - Melbourne, Victoria
  - Reservoir
- Bulgaria (10):
  - Burgas
  - Dobrich
  - Gabrovo
  - Karlovo
  - Lovech
  - Montana
  - Pazardzhik
  - Sofia
  - Stara Zagora
  - Veliko Tarnovo
- France (5):
  - Brest
  - Grenoble
  - Limoges Cedex1
  - Pierre-Bénite
  - Valenciennes
- Germany (7):
  - Pirmasens, Baden-Wurttemberg
  - Villingen-Schwenningen, Baden-Wurttemberg
  - Bonn, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Halle, Saxony-Anhalt
  - Berlin
  - Wuppertal
- Hungary (7):
  - Baja
  - Budapest
  - Debrecen
  - Esztergom
  - Kaposvár
  - Pécs
  - Szigetvár
- Israel (5):
  - Ashkelon
  - Hadera
  - Jerusalem
  - Kfar Saba
  - Nahariya
- Italy (9):
  - Chieti, Abruzzo
  - Napoli, Campania
  - Modena, Emilia-Romagna
  - Brescia, Lombardy
  - Cremona, Lombardy
  - Lecco, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - Livorno, Tuscany
- Japan (12):
  - Kitakyushu, Fukuoka
  - Ōkawa, Fukuoka
  - Muroran, Hokkaido
  - Hakusan, Ishikawa-ken
  - Morioka, Iwate
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Kuwana, Mie-ken
  - Chiba
  - Fukuoka
  - Nagano
  - Nara
- Poland (5):
  - Bialystok
  - Poznan
  - Radom
  - Szczecin
  - Żyrardów
- Romania (5):
  - Brasov
  - Bucharest
  - Constanța
  - Oradea
  - Târgu Mureş
- South Korea (2):
  - Bucheon-si, Gyeonggido
  - Seoul
- Spain (7):
  - Santiago de Compostela, A Coruña
  - L'Hospitalet de Llobregat, Barcelona
  - San Sebastián de los Reyes, Madrid
  - Alicante
  - Barcelona
  - Córdoba
  - Madrid
- Turkey (Türkiye) (3):
  - Ankara Univ. Medical Faculty, Ankara
  - Baskent University Medical Faculty, Ankara
  - Sifa University Medical Faculty, Izmir
- United Kingdom (13):
  - Reading, Berkshire
  - Cambridge, Cambridgeshire
  - Dundee, Dundee City
  - Brighton, East Sussex
  - Salford, Manchester
  - Hexham, Northumberland
  - Doncaster, South Yorkshire
  - Leeds, West Yorkshire
  - Chorley
  - Glasgow
  - Liverpool
  - London
  - Manchester

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/